CLINICAL TRIAL: NCT01766531
Title: Evaluation of Nutritional Status in ICU : Interest for the Measurement of Body Composition by Body Bioelectrical Impedance and Comparison With Several Methods
Acronym: IMPREA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Center of study in Human Nutrition, INRA, Department of Clinical Nutrition (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHU-0135
Record Dates: First submitted 2013-01-10; First posted 2013-01-11 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-11

CONDITIONS: Body Composition
Keywords: Bioelectrical impedance; Nutrition; Phase angle; ICU patients

ARMS (1):
- Body bioelectrical impedance (Experimental): comparison with four methods for assessing nutritional status. ; compare length of mechanical ventilation, length in ICU and energy expenditure rest between malnourished and non-malnourished patient
  Interventions: Device: body bioelectrical impedance

INTERVENTIONS:
Device: body bioelectrical impedance

SUMMARY:
Prospective cohort, monocentric non-randomized and interventional clinical study in ICU assessing the evolution of body composition using bioelectrical impedance analysis.

DETAILED DESCRIPTION:
Prospective, monocentric non-randomized and interventional clinical study in ICU assessing the evolution of body composition using bioelectrical impedance analysis (phase angle, fat mass, muscle mass, fat-free mass, body water); comparison with four methods for assessing nutritional status. ; compare length of mechanical ventilation, length in ICU and energy expenditure rest between malnourished and non-malnourished patient.

ELIGIBILITY:
Inclusion Criteria:

* ICU patients
* Written informed consent
* Adult patient

Exclusion Criteria:

* Pregnant patient
* Cardiac -pacemaker

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2012-06; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Evolution of fat-free mass | From day 4 to day 7
Evolution of fat-free mass | from day 8 to day 14
Evolution of fat-free mass | from day 14 to day 28

SECONDARY OUTCOMES:
Performance of the impedance to measure body evolution | in the first three days, from day 4 to day 7, from day 8 to day 14, from day 14 to day 28
Evolution of phase angle using bioelectrical impedance analysis | in the first three days, from day 4 to day 7, from day 8 to day 14, from day 14 to day 28
Comparison with four methods for assessing nutritional status | in the first three days, from day 4 to day 7, from day 8 to day 14, from day 14 to day 28
Compare length of mecanical ventilation, length in ICU and energy expenditure rest between malnourished ans non-malnourished patient | in the first three days, from day 4 to day 7, from day 8 to day 14, from day 14 to day 28

CONTACTS AND LOCATIONS:
Overall Officials: Sébastien PERBET, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France